CLINICAL TRIAL: NCT07022743
Title: Improving Treatment Outcomes in Chronic Myeloid Leukaemia Patients Using Imatinib and Artesunate Combination Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Famurewa Oluwatoyin, Mrs., Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMART Trial; IRB/IEC/Z0004553 (Other: Obafemi Awolowo University Teaching Hospital Complex Nigeria)
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: IMART Trial; Imatinib and artesunate; Chronic myeloid leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Artesunate

STUDY DESIGN:
Intervention Model Description: Group A: Imatinib naive patients placed on Imatinib alone Group B: Imatinib naive patients placed on Imatinib and artesunate Group C: Patients with sub-optimal response to imatinib placed on Imatinib and artesunate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Imatinib alone in newly diagnosed CML patients (Active Comparator): Imatinib (Glivec) at a dose of 400mg to newly diagnosed CML patients
  Interventions: Drug: Imatinib
- Group B: Imatinib and artesunate combination therapy (Experimental): Imatinib (Glivec) at a dose of 400mg daily and artesunate at a dose of 4mg/kg (not exceeding 200mg) daily in newly diagnosed CML patients
  Interventions: Drug: Imatinib; Drug: Artesunate
- Group C: Imatinib and artesunate in CML patients (Experimental): Imatinib (Glivec) 400mg and artesunate 400mg in CML patients with documented sub-optimal response to Imatinib, patients will be monitored monthly and reviewed after 3 months
  Interventions: Drug: Imatinib; Drug: Artesunate

INTERVENTIONS:
Drug: Imatinib — Imatinib is a first-line tyrosine kinase inhibitor which is used in the management of chronic myeloid leukaemia. It will be used by all the patients in the 3 arms of the study (Groups A, B and C)
  Other Names: Glivec
Drug: Artesunate — Artesunate has been established to reverse resistance to some chemotherapeutic agents. patients in 2 arms of the study (Groups B and C) will be given artesunate at 4mg/kg (not exceeding 200mg daily) in combination with imatinib
  Other Names: Tab Artesunate 50mg
  Arms: Group B: Imatinib and artesunate combination therapy; Group C: Imatinib and artesunate in CML patients

SUMMARY:
Chronic myeloid leukaemia (CML) is a blood cancer with an annual worldwide incidence of 1/100,000 population. Imatinib is used for the treatment of CML and has significantly improved the management of the disease. However, the incidence of treatment failure due to imatinib resistance has become a considerable burden (Sherbenou et al., 2007). Artesunate, an antimalarial drug, is reported to have anti-neoplastic effect either singly or in synergy with already established anti-neoplastic agents (Krishna et al., 2015).

The aim of the study is to evaluate the clinical effectiveness of an Imatinib-artesunate combination compared to imatinib alone and its possibility as an alternative option in the management of sub-optimal response in CML patients especially in low- and middle- income country like Nigeria where second line tyrosine kinase inhibitor may be out of reach.

The specific objectives are to:

1. Assess the safety of artesunate use beyond its traditional antimalarial dosing period in CML patients.
2. Compare treatment outcomes between patients on imatinib alone and patients on imatinib plus artesunate at 3, 6 and 12-months of follow-up.
3. Determine the effect of imatinib and artesunate combination on the achievement of major molecular remission in CML patients with sub-optimal response to imatinib.
4. Determine the effect of artesunate on imatinib pharmacokinetics following co-administration of the two drugs.

The main questions it aims to answer is:

* Does the use of artesunate in combination with imatinib in newly diagnosed CML patient give a better therapeutic outcome than using imatinib alone?
* Does combining artesunate with imatinib in CML patients with sub-optimal response to imatinib improve patients' response to imatinib?
* Does combining artesunate with imatinib in CML patients affect the pharmacokinetic parameter of imatinib?
* Is it safe to take artesunate at 4mg/day (not exceeding 200mg/day) for a 14day cycle in CML patients as demonstrated in other forms of cancer?

Participants will be assigned to one of the groups of the study and continue imatinib medication irrespective of the group assigned and come to clinic once a month for follow-up. Clinic visits will be immediately after a cycle of artesunate for groups B and C.

DETAILED DESCRIPTION:
Improving treatment outcomes in chronic myeloid leukaemia patients using Imatinib and Artesunate combination therapy.

Statement of Research Problem:

Imatinib is a first-line tyrosine kinase inhibitor (TKI) in the management of CML patients. At present, over one thousand Nigerians with CML are accessing free imatinib on the Glivec International Patient Assistance Program (GIPAP) platform at the Obafemi Awolowo University Teaching Hospital (OAUTH), Ile-Ife, Nigeria. This is the one of the two centres providing this service in the country and has been providing this service since 2003. However, only 40% of the patients had optimal clinical response while the rest had suboptimal response or treatment failure (Oyekunle et al., 2015). The high cost of alternative TKIs and/or stem cell transplantation hugely limits the treatment options available for Nigerian CML patients. Therefore, there is a strong need for an alternative therapeutic option that could optimize the management and clinical outcomes of CML in Nigeria and other resource-challenged countries.

Conceptual Framework of the Study:

This study explores drug repurposing for artesunate by investigating its anti-neoplastic effect in CML patients. Artesunate is a first-line antimalarial that has also demonstrated anti-leukemic activity in cell lines and murine models. Artesunate will be combined with imatinib and the synergy will be explored based on the multi-dimensional synergy of combination theory as described by Wooten (Wooten et al., 2019). The focus will be to evaluate the synergistic potency and synergistic efficacy of the combination. Synergistic potency is the amount of the change in drug potency, owing to the presence of another drug while synergistic efficacy is the percentage change in the maximal efficacy of the combination compared to the most efficacious single agent (Wooten et al., 2019). In this study, we will evaluate the pharmacokinetic interaction between artesunate and imatinib, and also determine the safety and efficacy of the combination, and the corresponding positive clinical outcomes in suboptimal CML patients. This approach has the potential to accelerate the translatability and reproducibility of this drug-synergy study by bridging the gap between the positive clinical outcome potential of the drug combination and the complexity of the study design.

Brief background:

CML is a clonal disease of the pluripotential haemopoietic stem cells, caused by a reciprocal translocation between chromosomes 9 and 22 with resultant formation of BCR-ABL1 chimeric gene and oncoprotein with constitutive tyrosine kinase activity. Through constitutive stimulation of multiple signal transduction pathways, this tyrosine kinase leads to neoplastic myeloid lineage expansion, primarily the granulocytic series but also megakaryocytic and only rarely, erythroid cells. Imatinib, is the first-line therapy for the management of Nigerian CML patients, which is consistent with the 2020 British Society of Haematology guidelines on the management of CML (Smith et al., 2020). Since 1998, when imatinib mesylate was first introduced, the treatment of CML has gained radical improvement with better outcome (Schmidli et al., 2005). Imatinib is available free of charge to patients in resource-limited countries such as Nigeria under the Glivec International Patient Assistance Program (GIPAP). A major limiting factor with this drug however, is the development of resistance which makes long-term disease-free remission difficult in some patients. The proportion of patients who achieved clinical cum molecular response after one year of standard dose imatinib daily ranged from 18% to 58% globally. In Nigeria, only 39.4% of CML patients on imatinib achieved major molecular response at ≥ 18 months of therapy while 25% of patients had imatinib-resistance from BCR-ABL1 kinase domain mutations which explained the cause of unsatisfactory response in this category of patients (Oyekunle et al., 2010). Lewandowski and colleagues (2009) also found twelve BCR-ABL mutations in 11 of 92 CML patients causing resistance to imatinib of which 40% were primary mutations while the rest 10.3% were secondary ones (Lewandowski et al., 2016).

Several alternative mechanisms aimed at overcoming imatinib resistance in CML patients have been explored. These include dose escalation of the drug or switching the patient to a second or third-line TKIs. The use of combinations of TKI and interferon [IFN] or pegylated interferon, omacetaxine mepussecinate have also been explored while allogeneic stem cell transplantation following failure of the novel TKIs has also been suggested to overcome the resistance. However, in a resource-limited setting, these options are not easily obtainable due to cost. The need therefore becomes inevitable to continuously search for an affordable alternative, which artesunate potentially presents.

Treatment milestones in Chronic Myeloid Leukaemia:

Mutations in the kinase domain of BCR-ABL are often responsible for resistance to imatinib. However, it is not necessary to request for mutation screening on a routine basis unless there is an indication for a loss of response (Sherbenou et al., 2007). The first therapeutic milestone is based on the evaluation after 3 months of therapy. It is expected that a complete haematologic response (CHR) is achieved at this time for an optimal response (Morotti et al., 2015). A partial haematological response (PHR) is considered a sub-optimal response according to the European Laeukaemia Net (ELN) recommendations (Hehlmann, 2020).

Artesunate use in Chronic Myeloid Leukaemia:

Artesunate is a semi-synthetic artemisinin compound and has been established to be the first-line treatment for malaria (Raffetin et al., 2018). However, it has been reported to possess anti-neoplastic effects either singly or in synergy with established anti-neoplastic drugs (Kumar et al., 2017). The mechanism of action is believed to be majorly due to endoperoxide-induced cytotoxicity via generation of reactive oxygen species when heam or ferrous iron activates the endoperoxide moiety of the drug, this effects toxicity to tumour cells via pathways involving growth arrest, reduced angiogenesis, DNA damage, and very importantly, apoptosis. There is however some evidence that artesunate possibly elicits its actions via multiple pathways including the regulation of key factors such as nuclear factor-kappa B [NFκ-B], BMI-1 and hypoxia-inducible factor-1ɑ pre-clinical study, using animal model of Xeno transplanted CML cells showed significant response to artesunate (Kim et al., 2015). Evidence of antitumor growth effect of this drug against urinary bladder and colorectal cancers has been demonstrated. The selective toxicity of artesunate to tumour cells is partly explained by reduced levels of antioxidant enzymes [e.g. catalase, glutathione peroxidase, superoxide dismutase] in these tumour cells (Krishna et al., 2015). Artesunate may also express toxicity towards some specific tumour proteins or biomarkers. Eling and co-researchers demonstrated this when they showed that artesunate selectively had high toxicity towards pancreatic ductal adenocarcinoma cells expressing KRas oncogene, but did not affect non-neoplastic human pancreatic ductal epithelial cells.

Artesunate at 200mg (2.2 - 3.9 mg/kg/day) for up to four weeks has been used as a continuous daily oral dose in colorectal and breast cancer patients without any significant toxicity. This dose was established to be safe and well tolerated over a four weeks period and is recommended for phase II/III trial. Chen et al recently showed that artesunate enhanced cancer cell death by inhibiting glycolysis in adriamycin-resistant chronic myeloid leukemia cells in vitro, thus giving credence to the molecular basis of artesunate in regulating glycolysis related enzymes (MDR1 and ABCG2) in leukemia cells. It is presently unknown whether artesunate can augment imatinib activity in the treatment of CML. The affordability and good clinical tolerability of artesunate and its proven anti-neoplastic property makes it suitable and worthwhile for this clinical trial in CML patients.

Details

1. . Study population: Consenting BCR-ABL positive chronic phase CML patients accessing imatinib at the OAUTHC, Nigeria.
2. . Study design: The study is a prospective randomized phase II clinical trial of artesunate and imatinib combination therapy in chronic phase CML patients. Patients will be recruited and followed up for at least 6 months of imatinib therapy.

   • Group C shall be 25 imatinib-exposed CML patients who have shown evidence of sub-optimal response to imatinib therapy. This group shall have standard-dose imatinib [400mg daily] plus artesunate [2mg/kg/day or 4mg/kg/day daily for 14 days every month]. Patients will be randomized to either doses called Group C2 or Group C4.

   Suboptimal response as defined by inability to achieve complete haematologic response (CHR) at 3months, major cytogenetic response (MCyR) at 6months, complete cytogenetic response (CCyR) at 12months or major molecular response (MMR) at 18months (Morotti et al., 2015).

   Group A: 25 newly diagnosed, imatinib naive, CP-CML patients placed on imatinib.

   Group B: 25 newly diagnosed, imatinib naive, CP-CML patients placed on imatinib and artesunate
3. . Sample Collections for pharmacokinetics analysis and imatinib levels 3mls of blood samples will be withdrawn from all the patients at pre-determined time intervals (0min, 30mins, 60mins, 120mins & 360mins) into EDTA tubes this will be further processed to obtain plasma and this will be stored at -20oC.
4. . Tests: The following investigations will be conducted at the time of recruitment and monthly; Full blood count, Renal function test, Liver function test, and Bcr-Abl testing (every three months).
5. . Pharmacokinetic analysis: A bio-analytical LC-MS/MS will be developed and validated according to ICH guidelines to simultaneously determine the amount of imatinib, its metabolite (N-desmethylimatinib) and artesunate and its metabolite (dihydroartemisin). This method will be used to quantify the amount of these drugs in the plasma of the patients at 3months, 6months and 12months of follow-up.
6. . Study End points: The primary endpoint will be the achievement of Major Molecular remission (MMR/MR3) with bcr/abl-1 gene transcript ≤0.1 and deep molecular response (MR4) with bcr/abl-1 gene transcript ≤0.01 at 12 months. The secondary endpoints will include plasma imatinib levels at 6 and 12 months, disease progression and adverse events relating to long-term use of artesunate.

(h). Statistical analysis: The cumulative incidence of molecular response rate at 12 months, the primary end point, will be estimated using the Kaplan-Meier method. Secondary endpoints regarding patient characteristics and safety indices will be estimated with the use of paired-sample tests. Confidence intervals will be estimated at the 95% confidence level and 2-sided P <0.05 will be considered to indicate statistical significance.

POTENTIAL VALUE OF THE RESEARCH RESULTS:

The results of the research may demonstrate if the use of artesunate is safe in CML patients beyond the traditional antimalaria dosing period as it has been determined in colorectal and breast cancer. The research may also evaluate if the combination of artesunate with imatinib may lead to better therapeutic outcome of the achievement of major molecular remission (MMR) in chronic phase CML patients and in the sub-optimal imatinib group. Also, it may show the influence of artesunate on the exposure of imatinib following co-administration of both.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed chronic phase CML patients
* Patients with sub-optimal response to imatinib therapy
* Ages between 18 years and 85 years with written informed consent

Exclusion Criteria:

* Patients with documented hypersensitivity to artesunate
* Patients with cardiovascular disease, pregnancy and inability to give consent will be excluded.
* Patients currently on any medication(s) that may interact with imatinib or affect its pharmacokinetics parameters (like rifampicin and ketoconazole) will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major molecular remission | 12 months
  The primary endpoint will be the achievement of Major Molecular remission (MMR/MR3) with bcr/abl-1 gene transcript ≤0.1 and deep molecular response (MR4) with bcr/abl-1 gene transcript ≤0.01 at 12 months.

SECONDARY OUTCOMES:
Plasma Imatinib levels | 3 months, 6 months and 12 months
  The outcome measure will be plasma imatinib levels within therapeutic window
Disease progression | 3 months, 6 months, 12 months
  The outcome measure will be the achievement of the expected treatment outcomes at 3, 6 and 12 months
Adverse events relating to long-term use of artesunate | Accessed after each cycle every month through the 12 months follow-up
  The outcome measure will be absence of any serious adverse event relating to long-term use of artesunate

CONTACTS AND LOCATIONS:
Overall Officials: Prof. R. A. Bolarinwa, Study Director — Obafemi Awolowo University, Ile-Ife; Dr. B. A. Adeagbo, Study Chair — Obafemi Awolowo University, Ile-Ife
Locations (1):
- Obafemi Awolowo University Teaching Hospital Complex, Ile-Ife, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No
The IPD might only be available to the principal investigator and study director and chair while the organized data and interpreted data and conclusions will be made available to the entire science community when the trial is concluded.

REFERENCES:
- [Background] Bethell D, Se Y, Lon C, Socheat D, Saunders D, Teja-Isavadharm P, Khemawoot P, Darapiseth S, Lin J, Sriwichai S, Kuntawungin W, Surasri S, Lee SJ, Sarim S, Tyner S, Smith B, Fukuda MM. Dose-dependent risk of neutropenia after 7-day courses of artesunate monotherapy in Cambodian patients with acute Plasmodium falciparum malaria. Clin Infect Dis. 2010 Dec 15;51(12):e105-14. doi: 10.1086/657402. Epub 2010 Nov 11. PMID 21070142
- [Background] Krishna S, Ganapathi S, Ster IC, Saeed ME, Cowan M, Finlayson C, Kovacsevics H, Jansen H, Kremsner PG, Efferth T, Kumar D. A Randomised, Double Blind, Placebo-Controlled Pilot Study of Oral Artesunate Therapy for Colorectal Cancer. EBioMedicine. 2014 Nov 15;2(1):82-90. doi: 10.1016/j.ebiom.2014.11.010. eCollection 2015 Jan. PMID 26137537
- [Background] White WL. Erratum to: Why I hate the index finger. Hand (N Y). 2011 Jun;6(2):233. doi: 10.1007/s11552-011-9321-0. Epub 2011 Mar 18. PMID 21776199
- [Background] Kim C, Lee JH, Kim SH, Sethi G, Ahn KS. Artesunate suppresses tumor growth and induces apoptosis through the modulation of multiple oncogenic cascades in a chronic myeloid leukemia xenograft mouse model. Oncotarget. 2015 Feb 28;6(6):4020-35. doi: 10.18632/oncotarget.3004. PMID 25738364
- [Background] Mander AP, Thompson SG. Two-stage designs optimal under the alternative hypothesis for phase II cancer clinical trials. Contemp Clin Trials. 2010 Nov;31(6):572-8. doi: 10.1016/j.cct.2010.07.008. Epub 2010 Aug 1. PMID 20678585
- [Background] Smith G, Apperley J, Milojkovic D, Cross NCP, Foroni L, Byrne J, Goringe A, Rao A, Khorashad J, de Lavallade H, Mead AJ, Osborne W, Plummer C, Jones G, Copland M; British Society for Haematology. A British Society for Haematology Guideline on the diagnosis and management of chronic myeloid leukaemia. Br J Haematol. 2020 Oct;191(2):171-193. doi: 10.1111/bjh.16971. Epub 2020 Jul 30. No abstract available. PMID 32734668
- [Background] Oyekunle AA, Bolarinwa RA, Oyelese AT, Salawu L, Durosinmi MA. Determinants of Overall and Progression-Free Survival of Nigerian Patients with Philadelphia-Positive Chronic Myeloid Leukemia. Adv Hematol. 2015;2015:908708. doi: 10.1155/2015/908708. Epub 2015 Sep 7. PMID 26435715
- [Background] Morotti A, Fava C, Saglio G. Milestones and monitoring. Curr Hematol Malig Rep. 2015 Jun;10(2):167-72. doi: 10.1007/s11899-015-0258-1. PMID 25921389

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT07022743/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT07022743/ICF_001.pdf